CLINICAL TRIAL: NCT01293461
Title: A Randomized, Blinded, Placebo-Controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of CBX129801 (Long-Acting Synthetic C-Peptide) After Subcutaneous Administration in Patients With Type 1 Diabetes Mellitus
Brief Title: Safety and Pharmacokinetics of CBX129801 in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cebix Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBX129801-PK-101
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Type 1 Diabetes; Diabetes Mellitus; Peripheral Diabetic Neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — CBX129801

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBX129801 (Experimental)
  Interventions: Drug: CBX129801
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBX129801 — Subcutaneous injection
  Arms: CBX129801
Drug: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess safety and tolerability and determine the pharmacokinetics of subcutaneous single and multiple (up to 12) dose administration of CBX129801 (long-acting synthetic C-peptide) in type 1 diabetes patients.

DETAILED DESCRIPTION:
This study will be conducted in two parts (Part 1 and Part 2). Part 1 will be conducted in three sequential dose cohorts with dose level escalated for each successive cohort. In Part 2 of the study, a dose regimen determined from the pharmacokinetic data from Part 1 will be administered in up to 40 additional subjects to achieve a target plasma concentration range that represents the most commonly observed physiological C-peptide levels in healthy, non-diabetic individuals.

ELIGIBILITY:
Key Inclusion Criteria:

* Give informed consent
* Aged 18 to 55 years (Part 1), Ages 18 to 65 years (Part 2)
* Stable type 1 diabetes mellitus (T1DM) for a minimum of 5 years
* Body mass index of 18-35 kg/m2
* Be C-peptide deficient (assessed by fasting concentration level)
* Normal renal function (assessed by serum creatinine)
* Be in good general health (besides T1DM)
* Have abnormal sural nerve conduction velocity observed bilaterally (Part 2 only)

Key Exclusion Criteria:

* Any significant cardiovascular, hematological, renal, hepatic, pulmonary, endocrine (except for diabetes mellitus), central nervous, or gastrointestinal condition or disease
* Unstable glucose control
* Have had a islet cell, kidney, and/or pancreas transplant
* Blood loss or blood donation within 56 days
* Drug or alcohol abuse (within 2 years) or recreational drug use (within 3 months)
* History or positive test result for Hepatitis B, C, and/or HIV
* Treatment with medication for peripheral neuropathy within 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To assess the single and multiple dose pharmacokinetics of plasma CBX129801 after subcutaneous (SC) administration of CBX129801 by estimating parameters of Cmax, Tmax, Cmin, AUClast, AUCinf, Tlag, Cav, CL/F, Vz/F, and half life. | For duration of study / 16 months
  Plasma CBX129801 will be used to assess the concentration versus time profiles and PK of CBX129801.
To assess the safety and tolerability of CBX129801 when administered SC by adverse events, injection site assessments, clinical laboratory tests, vital signs, physical examinations, and electrocardiograms. | For duration of study / 16 months

SECONDARY OUTCOMES:
To evaluate the technique of sensory nerve conduction velocity (SNCV) in the sural nerves in patients with type 1 diabetes mellitus. | Predose and 6 and 12 weeks postdose
To assess the immunogenicity of CBX129801 by occurrence of anti-CBX129801 antibody formation. | For duration of study / 16 months
To evaluate the technique of motor nerve conduction velocity (MNCV) in the peroneal nerves in patients with type 1 diabetes mellitus. | Predose and 6 and 12 weeks postdose
To evaluate the technique of vibration perception threshold (VPT) in patients with type 1 diabetes (Part 2 only) | Predose and 12 weeks postdose

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Escondido, California
  - Tustin, California
  - Walnut Creek, California
  - Aurora, Colorado
  - Butte, Montana
  - San Antonio, Texas
  - Olympia, Washington
  - Renton, Washington